CLINICAL TRIAL: NCT06829290
Title: Influence of Sarcopenia on the Course of the Diseases - Measured Using Ultrasound and Biochemical Markers
Brief Title: Influence of Sarcopenia on the Course of the Diseases
Status: Recruiting | Type: Observational
Sponsor: Universitatsmedizin Mainz - 1. Medizinische Klinik (Other)
Responsible Party: Principal Investigator, Wolfgang Maximilian Kremer, senior physician, Universitatsmedizin Mainz - 1. Medizinische Klinik
Other Study IDs: 2024-17561
Record Dates: First submitted 2025-02-04; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Liver Cirrhosis; Cancer; Cachexia; Sarcopenia; Mechanical Ventilation
Keywords: sarcopenia; ultrasound
MeSH Terms: conditions — Liver Cirrhosis; Neoplasms; Cachexia; Sarcopenia | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples Without DNA — EDTA 7,5 ml
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Ultrasound — Sonographisch measurement of muscles Blood muscle markers

SUMMARY:
Frailty is a geriatric syndrome that primarily affects older patients, but also patients with severe illnesses. It is particularly common among oncology patients, but also among patients with gastrointestinal diseases such as liver cirrhosis or pancreatitis. Sarcopenia, a form of frailty, is defined as a loss of muscle quantity, quality and function. Currently, complex methods such as CT or bioimpedance measurement are available. However, simpler techniques such as ultrasound-based measurement could be alternatives, but still require further validation. In addition, serological muscle markers could support and simplify diagnostics.

The aim of this project is to be able to estimate the prognosis of patients at an early stage by measuring sarcopenia using ultrasound and biomarkers.

DETAILED DESCRIPTION:
Frailty is a well-known syndrome that has a negative impact on many diseases and the course of disease. Patients affected by frailty are particularly vulnerable due to their inadequate ability to deal with extrinsic and intrinsic stressors. The prevalence of frailty increases with age, affecting 15% of people over the age of 65 and 25% of people over the age of 80.

Frailty is the end result of an interplay between malnutrition, cognitive impairment and muscle wasting. Each of these factors can be further examined and measured, but they also influence each other. In particular, reduced muscle mass and muscle function have been associated with poor quality of life and a worse course of disease. Sarcopenia is therefore becoming an increasingly important factor in various disease patterns and should be monitored further. Muscle atrophy and sarcopenia have multifactorial causes. Physical inactivity, chronic inflammation associated with chronic diseases, and malnutrition are particularly important in this context. Cross-sectional measurement of several muscles at the level of the lumbar vertebrae (L3), normalized to body size, and dual X-ray absorptiometry are currently the most commonly used techniques for measuring sarcopenia. However, complex equipment and procedures are required for the measurements. Furthermore, radiological imaging is costly and causes radiation exposure. Therefore, attempts have been made in the past to simplify the measurements. Sonographic measurement is a practical alternative. Many different muscle groups are accessible to ultrasound. In particular, the thigh muscles and the psoas major muscle can be easily visualized using sonography. The sonographic assessment of the psoas muscle area index (PMAI) and the thigh muscle thickness index (TMTI) are approaches to bedside morphometry that we use primarily.

Currently, little is known about serological muscle parameters. Measurement in the blood would be more elegant than sonographic muscle measurement. This would save additional instrumental diagnostics and still provide an impression of the musculature and thus possibly of the patient's fitness. Various biomarkers come into question for this. In particular, markers of muscle protein synthesis such as activin A/B and myostatin have already been described in individual collectives. However, biomarkers require further research, especially in various disease entities.

The investigators expect sonographic and laboratory measurements of the musculature to provide a better assessment of prognosis, quality of life and functional results during therapy.

ELIGIBILITY:
Inclusion Criteria:

* oncological patient in the field of gastrointestinal tumors
* patients with liver cirrhosis
* patients attending the intensive care unit

Exclusion Criteria:

* patients incapable of consenting
* patients with congenital muscle diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: oncological patient in the field of gastrointestinal tumors patients with liver cirrhosis patients attending the intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Complication | From the date of enrollment until the date of first documented complication (decopmensation, hospitalisation, death) from any cause whichever came first, assessed up to two years
  Number of patients with decompensation of the underlying disease (e.g. liver cirrhosis: hyropic decompensation) or hospitalisation or death

CONTACTS AND LOCATIONS:
Locations (1):
- Universitatsmedizin Mainz, Mainz, Rhineland-Palatinate, Germany

IPD SHARING:
Plan to Share IPD: Undecided
We will make the data available accordingly in the context of publications.

REFERENCES:
- [Background] Lena A, Hadzibegovic S, von Haehling S, Springer J, Coats AJ, Anker MS. Sarcopenia and cachexia in chronic diseases: from mechanisms to treatment. Pol Arch Intern Med. 2021 Dec 22;131(12):16135. doi: 10.20452/pamw.16135. Epub 2021 Nov 15. PMID 34775741
- [Background] Kremer WM, Labenz C, Kuchen R, Sagoschen I, Bodenstein M, Schreiner O, Worns MA, Sivanathan V, Weinmann A, Galle PR, Sprinzl MF. Sonographic assessment of low muscle quantity identifies mortality risk during COVID-19: a prospective single-centre study. J Cachexia Sarcopenia Muscle. 2022 Feb;13(1):169-179. doi: 10.1002/jcsm.12862. Epub 2021 Dec 8. PMID 34881516
- [Background] Pinto Dos Santos D, Kloeckner R, Koch S, Hoppe-Lotichius M, Zoller D, Toenges G, Kremer WM, Zimmermann T, Mittler J, Lang H, Duber C, Galle PR, Weinmann A, Sprinzl MF. Sarcopenia as prognostic factor for survival after orthotopic liver transplantation. Eur J Gastroenterol Hepatol. 2020 May;32(5):626-634. doi: 10.1097/MEG.0000000000001552. PMID 31725030
- [Background] Zhang JX, Yan HT, Ding Y, Liu J, Liu S, Zu QQ, Shi HB. Low Psoas-Muscle index is associated with decreased survival in hepatocellular carcinoma treated with transarterial chemoembolization. Ann Med. 2022 Dec;54(1):1562-1569. doi: 10.1080/07853890.2022.2081872. PMID 35639492
- [Background] Hida T, Ando K, Kobayashi K, Ito K, Tsushima M, Kobayakawa T, Morozumi M, Tanaka S, Machino M, Ota K, Kanbara S, Ito S, Ishiguro N, Hasegawa Y, Imagama S. <Editors' Choice> Ultrasound measurement of thigh muscle thickness for assessment of sarcopenia. Nagoya J Med Sci. 2018 Nov;80(4):519-527. doi: 10.18999/nagjms.80.4.519. PMID 30587866
- [Background] Hari A, Berzigotti A, Stabuc B, Caglevic N. Muscle psoas indices measured by ultrasound in cirrhosis - Preliminary evaluation of sarcopenia assessment and prediction of liver decompensation and mortality. Dig Liver Dis. 2019 Nov;51(11):1502-1507. doi: 10.1016/j.dld.2019.08.017. Epub 2019 Sep 20. PMID 31547952
- [Background] Kobayashi K, Maruyama H, Kiyono S, Ogasawara S, Suzuki E, Ooka Y, Chiba T, Kato N, Yamaguchi T. Application of transcutaneous ultrasonography for the diagnosis of muscle mass loss in patients with liver cirrhosis. J Gastroenterol. 2018 May;53(5):652-659. doi: 10.1007/s00535-017-1378-2. Epub 2017 Aug 18. PMID 28821966
- [Background] Takai Y, Katsumata Y, Kawakami Y, Kanehisa H, Fukunaga T. Ultrasound method for estimating the cross-sectional area of the psoas major muscle. Med Sci Sports Exerc. 2011 Oct;43(10):2000-4. doi: 10.1249/MSS.0b013e31821994cb. PMID 21448087
- [Background] McLean RR, Shardell MD, Alley DE, Cawthon PM, Fragala MS, Harris TB, Kenny AM, Peters KW, Ferrucci L, Guralnik JM, Kritchevsky SB, Kiel DP, Vassileva MT, Xue QL, Perera S, Studenski SA, Dam TT. Criteria for clinically relevant weakness and low lean mass and their longitudinal association with incident mobility impairment and mortality: the foundation for the National Institutes of Health (FNIH) sarcopenia project. J Gerontol A Biol Sci Med Sci. 2014 May;69(5):576-83. doi: 10.1093/gerona/glu012. PMID 24737560
- [Background] Cawthon PM, Peters KW, Shardell MD, McLean RR, Dam TT, Kenny AM, Fragala MS, Harris TB, Kiel DP, Guralnik JM, Ferrucci L, Kritchevsky SB, Vassileva MT, Studenski SA, Alley DE. Cutpoints for low appendicular lean mass that identify older adults with clinically significant weakness. J Gerontol A Biol Sci Med Sci. 2014 May;69(5):567-75. doi: 10.1093/gerona/glu023. PMID 24737559
- [Background] Cruz-Jentoft AJ, Sayer AA. Sarcopenia. Lancet. 2019 Jun 29;393(10191):2636-2646. doi: 10.1016/S0140-6736(19)31138-9. Epub 2019 Jun 3. PMID 31171417
- [Background] Durand F, Buyse S, Francoz C, Laouenan C, Bruno O, Belghiti J, Moreau R, Vilgrain V, Valla D. Prognostic value of muscle atrophy in cirrhosis using psoas muscle thickness on computed tomography. J Hepatol. 2014 Jun;60(6):1151-7. doi: 10.1016/j.jhep.2014.02.026. Epub 2014 Mar 6. PMID 24607622
- [Background] Benz E, Trajanoska K, Lahousse L, Schoufour JD, Terzikhan N, De Roos E, de Jonge GB, Williams R, Franco OH, Brusselle G, Rivadeneira F. Sarcopenia in COPD: a systematic review and meta-analysis. Eur Respir Rev. 2019 Nov 13;28(154):190049. doi: 10.1183/16000617.0049-2019. Print 2019 Dec 31. PMID 31722892
- [Background] Shachar SS, Williams GR, Muss HB, Nishijima TF. Prognostic value of sarcopenia in adults with solid tumours: A meta-analysis and systematic review. Eur J Cancer. 2016 Apr;57:58-67. doi: 10.1016/j.ejca.2015.12.030. Epub 2016 Feb 13. PMID 26882087
- [Background] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jan 1;48(1):16-31. doi: 10.1093/ageing/afy169. PMID 30312372
- [Background] Cruz-Jentoft AJ, Baeyens JP, Bauer JM, Boirie Y, Cederholm T, Landi F, Martin FC, Michel JP, Rolland Y, Schneider SM, Topinkova E, Vandewoude M, Zamboni M; European Working Group on Sarcopenia in Older People. Sarcopenia: European consensus on definition and diagnosis: Report of the European Working Group on Sarcopenia in Older People. Age Ageing. 2010 Jul;39(4):412-23. doi: 10.1093/ageing/afq034. Epub 2010 Apr 13. PMID 20392703
- [Background] Beaudart C, Zaaria M, Pasleau F, Reginster JY, Bruyere O. Health Outcomes of Sarcopenia: A Systematic Review and Meta-Analysis. PLoS One. 2017 Jan 17;12(1):e0169548. doi: 10.1371/journal.pone.0169548. eCollection 2017. PMID 28095426
- [Background] Xue QL. The frailty syndrome: definition and natural history. Clin Geriatr Med. 2011 Feb;27(1):1-15. doi: 10.1016/j.cger.2010.08.009. PMID 21093718